CLINICAL TRIAL: NCT01431677
Title: Muscle Biopsies in Healthy Volunteers: a Pilot Study
Brief Title: Muscle Biopsies in Healthy Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 999910221; 10-AG-N221
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-07-29

CONDITIONS: Sarcopenia; Frailty; Aging
Keywords: Muscle; Biopsy; Energetics; Sarcopenia; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty

INTERVENTIONS:
Procedure: Muscle Biopsy

SUMMARY:
Background:

- In individuals as they age, changes in muscle tissue can significantly affect their muscle strength and exercise endurance. This process, known as sarcopenia, may lead to decreased mobility and physical weakness, which is what we in general refer to as frailty. The causes of sarcopenia and why it affects some individuals more than others are not known, but many factors influence muscle physiology and function, including metabolic, hormonal, environmental, and lifestyle factors. Researchers interested in identifying factors involved in the start and progression of sarcopenia need of samples of human muscle tissue and cells for laboratory investigations.

Objectives:

* To train researchers in the appropriate procedures for performing muscle biopsies and collecting, labeling, and storing the samples.
* Develop a data base of specific scientific studies evaluating the physiological and metabolic function of muscle that can be used in future studies.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests, and will schedule a date for the muscle biopsy.
* Participants will have a muscle biopsy, with tissue and cells taken from the upper part of the thigh. A local anesthetic will be given for the procedure. Participants will also provide a blood sample and have an electrocardiogram to evaluate heart function.
* Participants will have a followup visit 1 week after the biopsy visit to evaluate the healing process and provide any further treatment for the affected area, after which they may fully resume normal activities.

DETAILED DESCRIPTION:
An important concept in pathologic aging is that in some individuals muscle strength and exercise endurance are significantly decreased through both quantitative and qualitative changes in muscle tissue. This process, termed sarcopenia, leads to frailty, a syndrome characterized by decreased mobility, weakness, and a very poor prognosis for survival, although the causal pathway for this association is not known. The causes of sarcopenia and why it affects some individuals more than others is not known. This is a complicated scientific question because many factors influence muscle physiology and function, including metabolic, hormonal, environmental, life-style, co-morbid medical problems and their treatments, etc. The National Institute on Aging (NIA) has a long-standing interest in sarcopenia and frailty and has established a number of observational studies aimed at understanding the cause and course of these age-related conditions. It is our goal to try to identify factors involved in the initiation and progression of sarcopenia and frailty, and to develop therapies that can reverse or slow these processes. To identify molecular and genetic changes that are associated with sarcopenia, it is crucial that human muscle biopsy specimens be available for laboratory investigations. This proposal will enable the Clinical Research Branch (CRB) to set up this procedure on the NIA Clinical Research Unit located on the fifth floor at Harbor Hospital, and to hone the practical skills that will be needed for analyzing muscle tissue from individuals in observational and interventional clinical trials. The goal will be to become facile at performing muscle biopsies, collecting, labeling and storing the samples, and to ensure that all equipment and expertise required to efficiently perform the procedure are in place. 14 healthy volunteers will be accrued to the study, however after this, the protocol will be kept open for the purpose of training other physicians or nurse practitioners in the biopsy procedure.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers over the age of 18

Normal screening laboratory studies including CBC, chem. 12 panel, PT/PTT, INR, UA, EKG

Ability to provide informed consent

EXCLUSION CRITERIA:

No history of bleeding diathesis

Subject is not on heparin, coumadin, plavix, or other anticoagulant

Subjects taking aspirin or non-steroidal anti-inflammatory agents must stop these 7 days before the biopsy

No allergy to lidocaine or bupivacaine

Subject has no active infections or chronic skin conditions that prevent access to the biopsy area

Unable to provide informed consent

No antibiotics for the past week

Positive pregnancy test

Positive for HIV, and/or positive for hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05-17; Primary Completion 2014-06-16 (Actual); Study Completion 2014-07-29 (Actual)

PRIMARY OUTCOMES:
Performing muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bandeen-Roche K, Xue QL, Ferrucci L, Walston J, Guralnik JM, Chaves P, Zeger SL, Fried LP. Phenotype of frailty: characterization in the women's health and aging studies. J Gerontol A Biol Sci Med Sci. 2006 Mar;61(3):262-6. doi: 10.1093/gerona/61.3.262. PMID 16567375
- [Background] Baur JA, Pearson KJ, Price NL, Jamieson HA, Lerin C, Kalra A, Prabhu VV, Allard JS, Lopez-Lluch G, Lewis K, Pistell PJ, Poosala S, Becker KG, Boss O, Gwinn D, Wang M, Ramaswamy S, Fishbein KW, Spencer RG, Lakatta EG, Le Couteur D, Shaw RJ, Navas P, Puigserver P, Ingram DK, de Cabo R, Sinclair DA. Resveratrol improves health and survival of mice on a high-calorie diet. Nature. 2006 Nov 16;444(7117):337-42. doi: 10.1038/nature05354. Epub 2006 Nov 1. PMID 17086191
- [Background] Civitarese AE, Ukropcova B, Carling S, Hulver M, DeFronzo RA, Mandarino L, Ravussin E, Smith SR. Role of adiponectin in human skeletal muscle bioenergetics. Cell Metab. 2006 Jul;4(1):75-87. doi: 10.1016/j.cmet.2006.05.002. PMID 16814734